CLINICAL TRIAL: NCT01820000
Title: Prospective Study to Obtain Preliminary Data to Determine the Efficacy of Non Contrast DWI Imaging Compared to CMR-DE
Brief Title: Efficacy of Non Contrast DWI(Diffusion Weighted Imaging) Imaging Compared to DMR-DE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jadranka Stojanovska, M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00032804
Record Dates: First submitted 2013-02-05; First posted 2013-03-28 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Heart Attack
MeSH Terms: conditions — Myocardial Infarction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diffusion Weighted Imaging with MRI scans (Experimental): Subjects will undergo a MRI (magnetic resonance imaging) scan where DWI (diffusion weighted imaging) will be performed. Subjects will not receive contrast during this sequence, but will receive contrast as standard MRI protocol.
  Interventions: Procedure: Diffusion Weighted Imaging with MRI scans

INTERVENTIONS:
Procedure: Diffusion Weighted Imaging with MRI scans — Subjects will have an MRI(magnetic resonance imaging)performed. This sequence will take no longer than 10 to 15 minutes to complete. Only DWI (diffusion weighted imaging) will be added to the standard cardiac MR protocol for viability which requires contrast injection. DWI(diffusion weighted imaging) sequence does not require contrast injection.

SUMMARY:
Use of MRI and DWI to diagnose cardiac scarring after heart attack.

DETAILED DESCRIPTION:
To discover new information about MRI (magnetic resonance imaging) called DWI (diffusion weighted imaging) and its ability to diagnose cardiac scarring.

CMR-DE (cardiac MR with delayed contrast enhancement) evaluates if there has been scarring in the heart muscle following a heart attack.

Subjects are injected with a contrast medication that makes the scarring visible if present. To prove the efficacy of DWI (diffusion weighted imaging) to provide the same images that CMR-DE (cardiac magnetic resonance with delayed contrast enhancement) provides.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 21 years of age and older
* Healthy volunteers
* subjects with a prior history of heart attack and prior CMR-DE imaging.

Exclusion Criteria:

* Women who are pregnant
* Subjects with GFR < 60 ml/min/1.73m2
* Subjects with ICD
* Subjects with coronary stents incompatible with 3T

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-12; Primary Completion 2014-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
presence and apparent diffusion coefficient (ADC) quantification of scar on (DWI) diffusion weighted image | single occurance
  Confirm the efficacy of diffusion weighted imaging in providing imaging that shows cardiac scarring without the injection of contrast.

CONTACTS AND LOCATIONS:
Overall Officials: Jadranka Stojanovska, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No